CLINICAL TRIAL: NCT06385158
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Oral Dose Escalation of GS1-144 Tablets and the Effects of Food on the Pharmacokinetics of GS1-144 in a Chinese Population
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GenSci074-101
Record Dates: First submitted 2024-04-11; First posted 2024-04-25 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Vasomotor System; Labile; Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GS1-144 tablet (Experimental)
  Interventions: Drug: GS1-144 tablet
- placebo controlled study (Placebo Comparator)
  Interventions: Drug: GS1-144 tablet

INTERVENTIONS:
Drug: GS1-144 tablet — GS1-144 tablet is an NK3R antagonist.

SUMMARY:
A Phase I clinical study evaluating the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple oral dose escalation of GS1-144 tablets and the effects of food on the pharmacokinetics of GS1-144 in a Chinese population

DETAILED DESCRIPTION:
The primary purpose of this study is to assess the safety and tolerability of single ascending doses of GS1-144 in healthy participants in Part 1 and assessing the food effect in Part 2,and to assess the safety and tolerability of multiple ascending doses of GS1-144 in healthy postmenopausal female participants in Part 3.

ELIGIBILITY:
Inclusion Criteria:

At the time of signing the informed consent form (ICF):

Part 1and Part 2 only: healthy male and female subjects aged between 18 and 45 years inclusive; Part 3 only: healthy women aged between 40 and 65 years inclusive who have undergone natural menopause (natural menopause is defined as surgically sterile (hysterectomy, bilateral salpingectomy, tubal ligation or bilateral oophorectomy - verbal confirmation through medical history review acceptable) or postmenopausal (no menses for 12 months and confirmed by FSH level ≥40 mlU/mL);

* Body weight ≥ 50 kg (male), ≥ 45 kg (female) with a body mass index between 19.0 and 27.9 kg/m2 inclusive at screening
* From signing the ICF to 1 month (female subjects) /3 months (male subjects and their female partners) after the end of the study, no family planning and egg/sperm donation plans, and effective contraceptive methods (such as IUD, bilateral tubal/vasectomy, condom and safe period calculation, etc.) (applicable to Parts 1 and 2)' ' ● Volunteer to sign ICF and be able to understand and comply with the requirements of this study

Exclusion Criteria:

Any known allergy to the components or analogues of the investigational product, or those with an allergic constitution (such as allergy to two or more drugs or foods)；

* A history of currently suffering from any other cardiovascular, gastrointestinal, endocrine, hematological, hepatic, immunological, metabolic, urinary, pulmonary, neurological, dermatological, psychiatric, renal and/or other major diseases deemed clinically significant by the investigator;
* Known/confirmed history of malignancy；
* A history of epileptic seizure or increased risk of epileptic seizure, or subjects with a recent history (within six months prior to screening) of head trauma leading to loss of consciousness or concussion;
* A history of currently suffering from hypothalamic dysfunction;
* Significant acute/chronic infections within two weeks prior to dosing;
* Undergone major surgical procedures (such as coronary artery bypass grafting, organ resection, gynecological surgery, etc.) within six months prior to screening or plan to undergo any surgery during the trial;
* Participated in other clinical trials (except those who have not received any intervention) within 3 months prior to dosing, Or are participating in other clinical trials.
* Have lost or donated more than 400 mL of blood within 3 months prior to screening;
* Have taken any prescription/over-the-counter drugs or dietary supplements ,within 7 days prior to dosing or within 5 half-lives of the drug (whichever is longer);
* Clinically significant abnormalities on physical examination or genitourinary ultrasound at the time of screening;
* Clinically significant abnormalities in vital signs, where the criteria for clinically significant blood pressure abnormalities are defined as systolic blood pressure ≥ 140 mmHg or < 90 mmHg, and diastolic blood pressure ≥ 90 mmHg or < 60 mmHg;
* Prolonged QTcF interval in 12-lead ECG results (> 450 ms for males, > 470 ms for females) or clinically significant abnormalities in other 12-lead ECG parameters at screening;
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), gamma-glutamyltransferase (GGT), total bilirubin (TBIL), blood creatinine (CRE), blood urea nitrogen (BUN), or international normalized ratio (INR) higher than the upper limit of normal (ULN) at screening, that are considered as clinically significant abnormalities by the investigator;
* Part 3 only: abnormal sex hormone levels at screening that are considered clinically significant by the investigator;
* Clinically significant abnormalities in thyroid function, parathyroid function, and neck ultrasound results at screening;
* Women with positive pregnancy test result or those who are breastfeeding before dosing;
* Positive hepatitis C virus antibody (HCV Ab), positive human immunodeficiency virus antibody (HIV Ab) or positive hepatitis B surface antigen (HbsAg) result at screening;
* Unable to refrain from consuming grapefruit, pomelo, grapefruit juice, or pomelo juice from 7 days prior to dosing until the end of the study;
* Unable to refrain from consuming any foods or beverages containing caffeine or xanthine (such as coffee, strong tea, chocolate, etc.) from 7 days prior to dosing until the end of the study;
* Unable to abstain from smoking/using tobacco products from 7 days prior to dosing until the end of the study, or positive urine cotinine test result before dosing
* Unable to refrain from consuming alcohol from 7 days prior to dosing until the end of the study, or positive breath alcohol test result before dosing;
* Any history of narcotic use or drug abuse, or positive urine drug screening result before dosing;
* Any medical or other condition, in the opinion of the investigator, may affect the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Part 1:Number of Participants With Treatment -Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to Day 4
  Number of participants with TEAEs and SAEs will be reported
Part 2: Number of Participants With Treatment -Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs). | Up to Day 9;
  Number of participants with TEAEs and SAEs will be reported.
Part 3: Number of Participants With TEAEs and SAEs | Up to Day 12
  Number of female post-menopausal participants with TEAEs and SAEs will be reported.

SECONDARY OUTCOMES:
Part1,Part2 and Part3 AUC0-t- Area Under the Drug Concentration-time Curve From Time 0 to the Last Sample Collection Time t for GS1-144 | Part 1 Day 1- pre-dose and up to 72 hour post-dose; Part 2 Days 1 and 6-pre-dose and up to 72 hour post-dose, Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose,
  AUC0-t will be assessed and reported.
Part 1 , Part2 and Part 3: AUC0-infinity- Area Under the Drug Concentration-time Curve From 0 to Infinity for GS1-144 | Part 1 Day 1- pre-dose and up to 72 hour post-dose; Part 2 Days 1 and 6-pre-dose and up to 72 hour post-dose, Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose,
  AUC0-infinity will be assessed and reported.
Part 1, Part2 and Part 3: Cmax- Maximum Observed Plasma Concentration for GS1-144 | Part 1 Day 1- pre-dose and up to 72 hour post-dose; Part 2 Days 1 and 6-pre-dose and up to 72 hour post-dose, Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose,
  Cmax will be assessed and reported.
Part 1 Part2 and Part 3: Tmax- Time to Reach the Maximum Plasma Concentration (Cmax) for GS1-144 | Part 1 Day 1- pre-dose and up to 24 hour post-dose; Part 2 Days 1 and 7-pre-dose and up to 30 hour post-dose
  Tmax will be assessed and reported.
Part 1 Part2 and Part 3:: T1/2- Terminal Half-life for GS1-144 | Time Frame: Part 1 Day 1- pre-dose and up to 72 hour post-dose; Part 2 Days 1 and 6-pre-dose and up to 72 hour post-dose, Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  T1/2 will be assessed and reported.
Part 1 Part2 and Part 3: CL/F- Apparent Clearance for GS1-144 | Part 1 Day 1- pre-dose and up to 72 hour post-dose; Part 2 Days 1 and 6-pre-dose and up to 72 hour post-dose, Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  CL/F will be assessed and reported.
Part 1 Part2 and Part 3: Vd/F- Apparent Volume of Distribution for GS1-144 | Part 1 Day 1- pre-dose and up to 72 hour post-dose; Part 2 Days 1 and 6-pre-dose and up to 72 hour post-dose, Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  Vd/F will be assessed and reported.
Cmax,ss- Observed Maximum Concentration at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  Cmax at steady state will be assessed and reported.
Part 3: Cmin,ss- Observed Minimum Concentration at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  Cmin at steady state will be assessed and reported.
Part 3: Tmax,ss- Time of Cmax at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  Tmax at steady state will be assessed and reported.
Part 3: Cavg,ss- Average Concentration at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  Cavg at steady state will be assessed and reported.
Part 3: AUC0-τ- Area Under the Drug Concentration-time Curve During the Dosing Interval at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  AUC0-T at steady state will be assessed and reported.
Part 3: CLss/F- CL for Bioavailability at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 30 hour post-dose
  CL/F at steady state will be assessed and reported.
Part 3: T1/2,ss- Terminal Half-life at Steady State for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  T1/2 at steady state will be assessed and reported.
Part 3: Accumulation Ratio for GS1-144 | Part 3 Days 1 and 7-pre-dose and up to 72 hour post-dose
  Accumulation Ratio will be assessed and reported.
Part 1: Baseline and placebo-adjusted changes in ∆∆QTc and other ECG parameters after oral administration of GF1-144 in healthy subjects | Part 1 Day 1- pre-dose and up to 24 hour post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided